CLINICAL TRIAL: NCT06011122
Title: Analysis of Implant Placement of Patients With Distal Radius Fractures in Western Britain,
Brief Title: Analysis of Implant Placement in Patients With Distal Radius Fractures in Western Brittany (REDIRA)
Acronym: REDIRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0084 - REDIRA
Record Dates: First submitted 2022-01-07; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Distal Radius Fracture
Keywords: Distal Radius fracture; Volar plate; Plate design; Watershed line; Plate positioning
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Zimmer Biomet: Patients who were operated with a Zimmer Biomet plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate
- Newclip Technics: Patients who were operated with a Newclip Technics plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate
- Stryker: Patients who were operated with a Stryker plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate
- Medartis: Patients who were operated with a Medartis plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate
- Medartis Footprint: Patients who were operated with a Medartis Footprint plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate
- Synthes: Patients who were operated with a Synthes plate
  Interventions: Procedure: Distal radius fracture ORIF with a specific volar plate

INTERVENTIONS:
Procedure: Distal radius fracture ORIF with a specific volar plate — Patients who had a distal radius fracture were treated surgically : an ORIF was realised with a volar plate

SUMMARY:
The purpose of this study was to determine the impact of design on plate position at the level of the distal radius. Six anterior wrist plates design were analyzed relative to the watershed line using the Soong classification. A total of 2723 anterior locking plate fixation cases were analyzed and divided into six groups: Zimmer Biomet, Newclip Technics, Stryker, Synthes, Medartis and Medartis Footprint. The number of plates recorded as Soong grade 0+1 was determined for each design, then compared using the Marascuilo procedure. The Zimmer Biomet and Newclip plates were proximal to the Watershed line significantly more often than those by Synthes and Medartis Footprint. Plate position with the Medartis design was significantly more proximal to the Watershed line compared to its companion design, the Medartis Footprint plate. Plate design is a deciding factor when treating distal radial fractures, to avoid impingement when implant removal is not routinely planned.

DETAILED DESCRIPTION:
This is a retrospective multicenter study involving several orthopedic surgeons with a trauma surgery practice within the public hospital centers of the department of Finistère. These include the CHU de Brest - Brest University Hospital Center (La Cavale Blanche), the HIA Clermont-Tonnerre military hospital (Hôpital d'Instruction des Armées - Armed Forces Teaching Hospital), the CH des Pays de Morlaix, the CH de Landerneau Ferdinand Grall, the CH de Carhaix and the CH de Cornouaille Quimper Concarneau. This study was approved by the local ethics committee. Among the cited hospital centers, the CHU de Brest is a level 1 trauma center, the CH des pays de Morlaix, the HIA military hospital and the CH de Cornouaille are level 2 trauma centers and the CH de Landerneau and Carhaix are level 3 trauma centers.

ELIGIBILITY:
To be included, patients had to have a digital radiographic file that could be used for the Soong classification. Among the volar plate fixation cases retrieved from the databases, we excluded patients that were not treated with a locking plate and those with a lateral x-ray that could not be interpreted. The inclusion criteria for lateral radiographs were alignment of the radius, lunate, capitate and third metacarpal bones, combined with radial-ulnar overlap (the ulnar styloid process projecting into the middle of the ulnar head).

Exclusion criteria:

Patient refusal No postoperative radiograph N=40 Poor quality radiograph N=214

Ages: 14 Years to 102 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included all patients with an intra-articular or extra-articular distal radial fracture managed by Volar Locking Plate fixation.
Sampling Method: Non-Probability Sample
Enrollment: 2723 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Influence of plate design on positioning | Retrospective study on Xray during 45 days
  The primary aim of this study was to compare six different VLPs meant to be positioned proximal to the watershed line, using the Soong classification.
  We will assess the rate of plates positioned "Soong 0+1" for each plate design

SECONDARY OUTCOMES:
Epidemiology | Retrospective study on Xray during 45 days
  to study the epidemiology of VLP fixation, per year, as recorded by the department of Finistère (northwestern France).
  We will assess for every year between 2009 and 2020 the prevalence of distal fracture treated by the use of a volar plate.
Impact of fracture type on plate positioning | Retrospective study on Xray during 45 days
  determine whether the type of fracture has an impact on plate position as defined by the Soong classification. We will assess the rates of different types of fractures according to AO classification and the rate of plates "Soong 0+1" for each fracture type

CONTACTS AND LOCATIONS:
Overall Officials: Hoel Letissier, MD MSc, Principal Investigator — Brest UH
Locations (5):
- France (5):
  - HIA Brest, Brest
  - CHRU de brest, Brest
  - CH de Landerneau, Landerneau
  - CH des pays de Morlaix, Morlaix
  - CHIC de Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- See also: Jerrhag D, Englund M, Karlsson MK, Rosengren BE. Epidemiology and time trends of distal forearm fractures in adults - a study of 11.2 million person-years in Sweden. BMC Musculoskelet Disord — https://doi.org/10.1186/s12891-017-1596-z
- See also: The Epidemiology of Upper Extremity Fractures in the United States, 2009. J Orthop Trauma 2015;29:e242-244 — https://doi.org/10.1097/BOT.0000000000000312
- See also: Corsino CB, Reeves RA, Sieg RN. Distal Radius Fractures. StatPearls, Treasure Island (FL) — https://doi.org/10.2106/JBJS.G.01569
- See also: Fractures of the distal part of the radius. The evolution of practice over time. Where's the evidence? — https://doi.org/10.2106/JBJS.M.00860
- See also: Brehmer JL, Husband JB. Accelerated rehabilitation compared with a standard protocol after distal radial fractures treated with volar open reduction and internal fixation: a prospective, randomized, controlled study — https://doi.org/10.1016/j.injury.2017.10.010